CLINICAL TRIAL: NCT02253550
Title: A Phase 2, Open-Label Study to Investigate the Efficacy and Safety of an 8-Week and 12-Week Regimen of Simeprevir in Combination With Sofosbuvir in Treatment-Naïve or -Experienced Subjects With Chronic Genotype 4 Hepatitis C Virus Infection With and Without Cirrhosis
Brief Title: Simeprevir in Combination With Sofosbuvir in Treatment-Naïve or -Experienced Adults With Chronic Genotype 4 Hepatitis C Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peter J. Ruane, M.D. (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor-Investigator, Peter J. Ruane, M.D., Principal Investigator, President, Peter J. Ruane, M.D., Inc.
Organization: Peter J. Ruane, M.D., Inc. (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMC435HPC2012
Record Dates: First submitted 2014-09-17; First posted 2014-10-01 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Simeprevir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cirrhosis (Experimental): Patients with confirmed presence of cirrhosis will received 12 weeks of treatment with Sofosbuvir and Simeprevir
  Interventions: Drug: Simeprevir; Drug: Sofosbuvir
- Non-Cirrhotic (Experimental): Patients with confirmed absence of cirrhosis will received 8 weeks of treatment with Sofosbuvir and Simeprevir
  Interventions: Drug: Simeprevir; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Simeprevir — Simeprevir is a Hepatitis C Virus (HCV) NS3/4A protease inhibitor approved in the United States, Canada and Japan for the treatment of chronic HCV infection.
  Other Names: Olysio; TMC435
Drug: Sofosbuvir — Sofosbuvir is a nucleotide NS5B polymerase inhibitor developed by Gilead Sciences Inc. and approved for the treatment of chronic HCV infection.
  Other Names: Sovaldi; GS-7977; PSI-7977

SUMMARY:
This study will look at the safety and efficacy of 8 week and 12 week treatment with Sofosbuvir and Simeprevir in treatment-naïve and treatment-experienced patients with chronic hepatitis C genotype 4.

DETAILED DESCRIPTION:
Patients with confirmed absence of cirrhosis will receive 8 weeks of treatment with Sofosbuvir and Simeprevir. Patients with confirmed presence of cirrhosis will receive 12 weeks of treatment with Sofosbuvir and Simeprevir. All patients will followed for 24 weeks post-treatment. Presence or absence of cirrhosis will be evaluated by FibroScan if no historical liver biopsy or FibroScan is available.

ELIGIBILITY:
Inclusion Criteria:

* HCV genotype 4 infection
* HCV RNA >10,000 IU/mL at screening.

Exclusion Criteria:

* Evidence of clinical hepatic decompensation (history or current evidence of ascites, bleeding varices or hepatic encephalopathy).
* Any liver disease of non-HCV etiology. This includes, but is not limited to, acute hepatitis A, drug- or alcohol-related liver disease, autoimmune hepatitis, hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency, non-alcoholic steatohepatitis, primary biliary cirrhosis, or any other non-HCV liver disease considered clinically significant by the investigator.
* Infection/co-infection with HCV non-genotype 4.
* Co-infection with human immunodeficiency virus (HIV) type 1 or type 2 (HIV-1 or HIV-2) (positive HIV-1 or HIV-2 antibodies test at screening).
* Co-infection with hepatitis-B virus (hepatitis-B-surface-antigen [HBsAg] positive).
* Presence of significant co-morbidities or conditions that would compromise the subject's safety and could interfere with the subject's participation for the full duration of the study in the opinion of the investigator
* Previously been treated with any direct acting anti-HCV agent (approved or investigational) for chronic HCV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Sustained Virologic Response 12 Weeks after Treatment Completion (SVR12) | 12 weeks post-treatment
  HCV RNA will be measured 12 weeks post-treatment to evaluate SVR

SECONDARY OUTCOMES:
Sustained Virologic Response 4 and 24 Weeks after Treatment Completion | 4 and 24 weeks post-treatment
  HCV RNA will be measured 4 and 24 weeks post-treatment to evaluate SVR

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Ruane, MD, Principal Investigator — Peter J. Ruane, MD, Inc.
Locations (1):
- Peter J. Ruane, MD, Inc., Los Angeles, California, United States